CLINICAL TRIAL: NCT03466788
Title: Impact of Adjuvant Chemotherapy on the Quality of Life of Patients Treated for Stage II / III Endometrial Cancer
Acronym: EndoQOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EndoQOL
Record Dates: First submitted 2018-02-27; First posted 2018-03-15 (Actual); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Cancer; Chemotherapy Effect; Quality of Life
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Social Conditions

STUDY DESIGN:
Who Masked: Participant
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients treated with chemotherapy (Other)
  Interventions: Other: Self questionnaires of quality of life and living conditions
- Patients not treated with chemotherapy (Other)
  Interventions: Other: Self questionnaires of quality of life and living conditions

INTERVENTIONS:
Other: Self questionnaires of quality of life and living conditions — Patients will complete self-questionnaires of living conditions and quality of life (QLQ-C30; EN24; CIPN20; IPAQ; HADS)

SUMMARY:
Through this study, The investigator believe to evaluate the impact in terms of overall quality of life of adjuvant chemotherapy in patients with locally advanced endometrial cancer at a distance from their care

DETAILED DESCRIPTION:
Endometrial cancer is the fourth most common cancer in women in developed countries. The diagnosis is often made at a localized stage (67% of cases), making it a relatively good cancer prognosis with a 5-year all-stage survival of 81.7%.

Its management at the localized stage is based on surgery and radiotherapy. Adjuvant chemotherapy may be offered in addition to radiotherapy, but its place is still debated. It is classically delivered sequentially before or after radiotherapy, concomitant radiochemotherapy not being a standard. It is generally recommended in case of stage III, and for the earlier stages, its use is based on various prognostic factors (histological type, grade, emboli) and the feasibility of treatment (age, general condition, comorbidities). In fact, patients treated for endometrial cancer are elderly (median age 63 years) and in the majority of cases present comorbidities (diabetes, obesity and hypertension). Chemotherapy can induce side effects that can persist and potentially alter the quality of life of these often fragile patients. Although the impact of surgery and radiotherapy on the quality of life has been well studied, there is insufficient literature data for adjuvant chemotherapy. The investigator propose a case-control study that will evaluate the quality of life and late sequelae of patients treated for locally advanced endometrial cancer with sequential adjuvant chemotherapy before or after radiotherapy at a distance from their management. comparing their results to a group of patients who had been treated with postoperative radiotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

For all patients:

* Women over 18 years of age, with histologically confirmed histologic type 1 or type 2 endometrial adenocarcinoma, with FIGO postoperative II or III stage operated between 2011 and 2015, with at least 2 years of follow-up compared to the last course of chemotherapy;
* Recommended surgery such as hysterectomy and bilateral salpingo-oophorectomy, non-mandatory surgical nodal staging;
* Pelvic radiotherapy +/- lumbar-aortic irradiation, optional brachytherapy;
* No recurrence of endometrial cancer at baseline;
* Absence of evolutionary neurological antecedent (multiple sclerosis, neurodegenerative pathology ...);
* Absence of progressive psychiatric pathology (i.e. psychiatric hospitalization, bipolar disorder, schizophrenia, personality disorders ...);
* No opposition to the collection of data;
* Patient deemed fit to answer a written questionnaire.

For the patient in the chemotherapy group - Chemotherapy after surgery that can be performed before or after radiotherapy

Exclusion Criteria:

For all patients:

* Sarcoma or carcinosarcoma;
* Stage FIGO I or IV;
* Macroscopic tumor residue after surgery;
* Recurrence of endometrial cancer or diagnosis of any other cancerous pathology after diagnosis of endometrial cancer (except non-melanotic skin tumors with complete excision), within 5 years;
* drug use;
* Abuse of alcohol.

For the patient in the chemotherapy group

* Chemotherapy before surgery;
* Chemotherapy concomitant with radiotherapy

For the patient in the group without chemotherapy

- Chemotherapy whether before or after surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2020-03-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre François Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Gustave Roussy, Villejuif

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Treated With Chemotherapy: Case patients had sequential carboplatin AUC5 -paclitaxel 175 mg/m2 J1=J21, excluding concomitant chemotherapy with radiotherapy.
- Patients Not Treated With Chemotherapy: Control patients received only surgery and radiotherapy.
Period: Overall Study
Arm/Group | Patients Treated With Chemotherapy | Patients Not Treated With Chemotherapy
Started | 20 | 30
Completed | 20 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Treated With Chemotherapy | Patients Not Treated With Chemotherapy | Total
Number analyzed (Participants) | 20 | 30 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (9) | 69.6 (10) | 67.9 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants] — All patients are woman (ovarian cancer)
  Participants
    Female | 20 | 30 | 50
    Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
WHO performance status [Count of Participants; unit: Participants] — WHO performance status graded 0 "fully active, able to carry on all pre-disease performance without restriction", 1 "restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work", 2 "ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours", 3 "capable of only limited selfcare, confined to bed or chair more than 50% of waking hours", 4 "Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair", 5 "Dead".
  Participants
    0 | 16 | 24 | 40
    1 | 2 | 2 | 4
    2 | 1 | 0 | 1
    Unknown | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Impact in Terms of Overall Quality of Life of Adjuvant Chemotherapy by the QLQ-C30 Questionnaire
Description: The Quality of life questionnaire (QLQ-C30) contains 29 items dealing with fatigue, pain, nausea and vomiting, general condition and social, emotional and cognitive functions. It is currently used in many clinical trials in oncology. Here is the glodal health status scale of the QLQ-C30 questionnaire, ranging from 0 to 100, with high score indicating good quality of life.
Time Frame: 2 years after chemotherapy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients treated with chemotherapy | Patients not treated with chemotherapy
Number analyzed (Participants) | 20 | 30
units on a scale | 61.7 (13.2) | 71.1 (18.9)

2. Secondary Outcome: Neurotoxicity Induced by Adjuvant Chemotherapy by the CIPN20 Questionnaire
Description: The quality of life Questionnaire Chemotherapy Induced Peripheral Neuropathy (QLQ-CIPN20) is a questionnaire specifically dedicated to the evaluation of peripheral neuropathies induced by chemotherapy. This quality of life questionnaire is composed of 20 items from 0 to 4 and has been tested in a large international clinical trial. Here is the sensory scale, ranging from 0 to 100, with high scoring indicating high symptom of neuropathy
Time Frame: 2 years after chemotherapy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients treated with chemotherapy | Patients not treated with chemotherapy
Number analyzed (Participants) | 20 | 30
units on a scale | 20.04 (18.5) | 6.86 (11.2)

3. Secondary Outcome: Different Domains of Quality of Life Impacted Remotely by Chemotherapy by the QLQ-C30 Questionnaire
Description: The Quality of life questionnaire (QLQ-C30) contains 29 items dealing with fatigue, pain, nausea and vomiting, general condition and social, emotional and cognitive functions. QLQ-C30 scoring cinludes 5 functionning scales (physical, role, emotional, cognitive and social), ranging from 0 to 100, with high score indicating high level of quality-of-life.
  QLQ-C30 scoring includes 9 symptom scales (fatigue, nausea/vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhea and financial difficulties), ranging from 0 to 100, with high score indicating poor level of quality-of-life.
Time Frame: 2 years after chemotherapy
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Patients treated with chemotherapy | Patients not treated with chemotherapy
Number analyzed (Participants) | 20 | 30
points
  Physical functioning | 75.3 (19) | 76.8 (23)
  Role functioning | 77.2 (24.3) | 80.7 (27)
  Emotional functioning | 67.1 (27) | 79.5 (24.6)
  Cognitive functioning | 76.7 (21.9) | 81 (24.3)
  Social functioning | 75.4 (30.6) | 84.6 (24.9)
  Fatigue | 38.8 (23.8) | 22.7 (17.7)
  Nausea and vomiting | 5.8 (16.5) | 8.9 (24.7)
  Pain | 31.6 (33.7) | 25 (25.5)
  Dyspnea | 22.8 (25) | 16 (23.3)
  Insomnia | 36.8 (31.2) | 32.2 (24.4)
  Loss of appetite | 15 (27.5) | 7.1 (16.6)
  Financial difficulties | 18.3 (33.3) | 6 (15.9)
  Constipation | 30 (35.7) | 19.5 (31.5)
  Diarrhea | 13.3 (22.7) | 25.9 (35)

4. Other Pre Specified Outcome: Anxiety by the HADS Questionnaire
Description: The Hospital Anxiety and Depression Scale (HADS) It is a quick and easy self-questionnaire that assesses both anxious and depressive dimensions (7 items for each dimension). Here is the scale of Anxiety, ranging from 0 to 21, with high score reflecting high level of anxiety.
Time Frame: 2 years after chemotherapy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients treated with chemotherapy | Patients not treated with chemotherapy
Number analyzed (Participants) | 20 | 30
units on a scale | 9.7 (5.3) | 7.7 (4.9)

5. Other Pre Specified Outcome: Depression by the HADS Questionnaire
Description: The Hospital Anxiety and Depression Scale (HADS) It is a quick and easy self-questionnaire that assesses both anxious and depressive dimensions (7 items for each dimension). Here is the depression scale, ranging from 0 to 21, with high score indicating high level of depression.
Time Frame: 2 years after chemotherapy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients treated with chemotherapy | Patients not treated with chemotherapy
Number analyzed (Participants) | 20 | 30
units on a scale | 5.8 (4.2) | 4.9 (3.5)

ADVERSE EVENTS:
Time Frame: 2 years, assessed retrospectively. Patients were included 2 years after their treatment.
Arm/Group | Patients Treated With Chemotherapy | Patients Not Treated With Chemotherapy
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/30
Other Adverse Events (participants affected / at risk) | 16/20 | 25/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Treated With Chemotherapy (N=20) | Patients Not Treated With Chemotherapy (N=30)
DYSPNOEA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1) | 0 (0)
NEUROPATHY PERIPHERAL (NERVOUS SYSTEM DISORDERS) | 7 (7) | 0 (0)
NAUSEA (GASTROINTESTINAL DISORDERS) | 9 (9) | 2 (2)
POLLAKIURIA (RENAL AND URINARY DISORDERS) | 1 (1) | 2 (2)
DIARRHOEA (GASTROINTESTINAL DISORDERS) | 9 (9) | 13 (13)
RADIATION SKIN INJURY (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 0 (0) | 1 (1)
ABDOMINAL PAIN (GASTROINTESTINAL DISORDERS) | 1 (1) | 2 (2)
PLEURAL EFFUSION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1) | 0 (0)
CYSTITIS (INFECTIONS AND INFESTATIONS) | 4 (4) | 8 (8)
INTERMENSTRUAL BLEEDING (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 0 (0) | 1 (1)
VAGINAL INFECTION (INFECTIONS AND INFESTATIONS) | 0 (0) | 1 (1)
DYSPAREUNIA (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 0 (0) | 2 (2)
PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 1 (1)
RENAL FAILURE (RENAL AND URINARY DISORDERS) | 0 (0) | 1 (1)
ASTHENIA (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 3 (3) | 1 (1)
ANAEMIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 2 (2) | 0 (0)
LYMPHOEDEMA (VASCULAR DISORDERS) | 3 (3) | 0 (0)
RADIATION PROCTITIS (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 1 (1) | 0 (0)
FEBRILE BONE MARROW APLASIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 1 (1) | 0 (0)
URINARY INCONTINENCE (RENAL AND URINARY DISORDERS) | 0 (0) | 8 (8)
FATIGUE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 1 (1)
DEPRESSION (PSYCHIATRIC DISORDERS) | 1 (1) | 0 (0)
ARTHRALGIA (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1) | 0 (0)
VOMITING (GASTROINTESTINAL DISORDERS) | 2 (2) | 2 (2)
THROMBOCYTOPENIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 1 (1) | 0 (0)
PROCTITIS (GASTROINTESTINAL DISORDERS) | 1 (1) | 1 (1)
URINARY TRACT INFECTION (INFECTIONS AND INFESTATIONS) | 0 (0) | 1 (1)
PELVIC PAIN (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 0 (0) | 1 (1)
ANAL INFLAMMATION (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
HAEMORRHOIDS (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT03466788/Prot_000.pdf